CLINICAL TRIAL: NCT00441883
Title: A Phase 2, 28 Day Parallel-Group, Double-Masked, Dose-Finding Study Comparing the Safety and Efficacy of PF-03187207 to Latanoprost
Brief Title: Dose-Finding Study Comparing the Safety and Efficacy of Latanoprost to a Novel Treatment for Glaucoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Collaborators: NicOx Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: A9441001
Record Dates: First submitted 2007-02-27; First posted 2007-03-01 (Estimated); Results first posted 2020-08-27 (Actual); Last update posted 2020-09-14 (Actual); Status verified 2020-09

CONDITIONS: Primary Open Angle Glaucoma; Ocular Hypertension; Pigmentary Glaucoma; Pseudoexfoliative Glaucoma
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension | interventions — Latanoprost

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PF-03187207 and Latanoprost Vehicle (Experimental): One drop of each, once daily in study eye for 28 days
  Interventions: Drug: PF-03187207 and Latanoprost Vehicle
- Latanoprost 0.005% and PF-03187207 Vehicle (Active Comparator): One drop of each, once daily in study eye for 28 days
  Interventions: Drug: Latanoprost 0.005% and PF-03187207 Vehicle

INTERVENTIONS:
Drug: PF-03187207 and Latanoprost Vehicle
  Arms: PF-03187207 and Latanoprost Vehicle
Drug: Latanoprost 0.005% and PF-03187207 Vehicle
  Arms: Latanoprost 0.005% and PF-03187207 Vehicle

SUMMARY:
This study will evaluate the safety and efficacy of PF 03187207.

ELIGIBILITY:
Inclusion Criteria:

-Diagnosis of primary open angle glaucoma (including pigmentary or pseudoexfoliative) or ocular hypertension in one or both eyes

Exclusion Criteria:

-Closed or barely open anterior chamber angle or a history of acute angle closure in either eye

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Actual)
Dates: Start 2007-03; Primary Completion 2008-02 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Harper, Study Director — Bausch & Lomb Incorporated
Locations (18):
- United States (18):
  - Pfizer Investigational Site, Artesia, California
  - Pfizer Investigational Site, Newport Beach, California
  - Pfizer Investigational Site, Petaluma, California
  - Pfizer Investigational Site, Poway, California
  - Pfizer Investigational Site, Danbury, Connecticut
  - Pfizer Investigational Site, Jacksonville, Florida
  - Pfizer Investigational Site, Ormond Beach, Florida
  - Pfizer Investigational Site, Atlanta, Georgia
  - Pfizer Investigational Site, Evansville, Indiana
  - Pfizer Investigational Site, Louisville, Kentucky
  - Pfizer Investigational Site, Rochester, New York
  - Pfizer Investigational Site, Charlotte, North Carolina
  - Pfizer Investigational Site, High Point, North Carolina
  - Pfizer Investigational Site, Tulsa, Oklahoma
  - Pfizer Investigational Site, Cranberry Township, Pennsylvania
  - Pfizer Investigational Site, Pittsburgh, Pennsylvania
  - Pfizer Investigational Site, Memphis, Tennessee
  - Pfizer Investigational Site, Austin, Texas

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A9441001&StudyName=A%20Phase%202%2C%20Dose-Finding%20Study%20Comparing%20the%20Safety%20and%20Efficacy%20of%20Latanoprost%20to%20a%20Novel%20Treatment%20for%20Glaucoma

RESULTS

PARTICIPANT FLOW:
Groups:
- PF-03187207 0.024% AM: PF-03187207 0.024% dosed in the morning
- PF-03187207 0.040% AM: PF-03187207 0.040% dosed in the morning
- PF-03187207 0.040% PM: PF-03187207 0.040% dosed in the evening
- Latanoprost 0.005% AM: Latanoprost 0.005% dosed in the morning
- Latanoprost 0.005% PM: Latanoprost 0.005% dosed in the evening
Period: Overall Study
Arm/Group | PF-03187207 0.024% AM | PF-03187207 0.040% AM | PF-03187207 0.040% PM | Latanoprost 0.005% AM | Latanoprost 0.005% PM
Started | 43 | 32 | 28 | 28 | 45
ITT Population (Participants randomized and at least 1 dose of study medication; by randomized treatment.) | 43 | 30 | 30 | 30 | 43
Per Protocol Population (Participant randomized with no major protocol violations; by treatment received.) | 38 | 29 | 25 | 24 | 38
Safety Population (Participants randomized with at least 1 dose of study medication; by treatment received.) | 43 | 32 | 28 | 28 | 45
Completed | 42 | 32 | 28 | 28 | 43
Not Completed | 1 | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: ITT population
Groups:
- Total: Total of all reporting groups
Arm/Group | PF-03187207 0.024% AM | PF-03187207 0.040% AM | PF-03187207 0.040% PM | Latanoprost 0.005% AM | Latanoprost 0.005% PM | Total
Number analyzed (Participants) | 43 | 30 | 30 | 30 | 43 | 176
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.1 (10.2) | 61.9 (10.9) | 61.8 (9.0) | 62.1 (11.3) | 63.6 (12.8) | 63.4 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 21 | 20 | 23 | 27 | 118
  Male | 16 | 9 | 10 | 7 | 16 | 58

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline Mean Diurnal Intraocular Pressure (IOP) in the Study Eye on Day 28
Description: Intraocular pressure (IOP) was measured using a Goldmann applanation tonometer. Diurnal IOP, defined as the mean IOP over the day based on values obtained at 8 AM, 10 AM, 1 PM, and 4 PM, was calculated for each visit. Both eyes were tested, with the right eye preceding the left eye. The operator initially set the dial at 10 mmHg, then looked through the slit lamp and adjusted the dial to take the reading, and then recorded the results. The procedure was repeated on the same eye twice consecutively. If the measurements were within 2 mmHg or less of each other, the mean of the 2 readings was recorded as the IOP at that time point. If the 2 readings were more than 2 mmHg of each other, a third (consecutive) reading was taken and the median (middle) IOP was recorded as the IOP at that time point.
Time Frame: Baseline, 28 days
Population: Per protocol population
Measure: Mean (Standard Deviation); unit: mmHg (milimeters of mercury)
Arm/Group | PF-03187207 0.024% AM | PF-03187207 0.040% AM | PF-03187207 0.040% PM | Latanoprost 0.005% AM | Latanoprost 0.005% PM
Number analyzed (Participants) | 38 | 29 | 25 | 24 | 38
mmHg (milimeters of mercury) | -6.96 (2.772) | -7.09 (2.123) | -8.20 (4.011) | -6.02 (2.322) | -7.28 (2.871)

2. Secondary Outcome: Change From Baseline in Mean Intraocular Pressure IOP at the Day 7, 14, and 21 Visits
Description: Intraocular pressure (IOP) was measured using a Goldmann applanation tonometer. gBoth eyes were tested, with the right eye preceding the left eye. The operator initially set the dial at 10 mmHg, then looked through the slit lamp and adjusted the dial to take the reading, and then recorded the results. The procedure was repeated on the same eye twice consecutively. If the measurements were within 2 mmHg or less of each other, the mean of the 2 readings was recorded as the IOP at that time point. If the 2 readings were more than 2 mmHg of each other, a third (consecutive) reading was taken and the median (middle) IOP was recorded as the IOP at that time point.
Time Frame: Baseline, Day 7, Day 14, and Day 21
Population: Per protocol population
Measure: Mean (Standard Deviation); unit: mmHg (milimeters of mercury)
Arm/Group | PF-03187207 0.024% AM | PF-03187207 0.040% AM | PF-03187207 0.040% PM | Latanoprost 0.005% AM | Latanoprost 0.005% PM
Number analyzed (Participants) | 38 | 29 | 25 | 24 | 38
mmHg (milimeters of mercury)
  Day 7 | -6.58 (2.630) | -7.20 (2.555) | -7.85 (3.970) | -5.49 (1.926) | -6.82 (2.556)
  Day 14 | -7.20 (2.776) | -7.20 (2.595) | -8.18 (3.267) | -5.27 (2.679) | -7.0 (2.295)
  Day 21 | -6.68 (2.133) | -7.34 (2.579) | -8.35 (3.309) | -5.81 (2.625) | -7.04 (2.640)

3. Secondary Outcome: Percentage of Participants With Intraocular Pressure (IOP) Less Than or Equal to 18 mmHg at Any Visit Through Day 28
Description: Intraocular pressure (IOP) was measured using a Goldmann applanation tonometer. Both eyes were tested, with the right eye preceding the left eye. The operator initially set the dial at 10 mmHg, then looked through the slit lamp and adjusted the dial to take the reading, and then recorded the results. The procedure was repeated on the same eye twice consecutively. If the measurements were within 2 mmHg or less of each other, the mean of the 2 readings was recorded as the IOP at that time point. If the 2 readings were more than 2 mmHg of each other, a third (consecutive) reading was taken and the median (middle) IOP was recorded as the IOP at that time point.
Time Frame: 28 days
Population: Per protocol population
Measure: Count of Participants; unit: Participants
Arm/Group | PF-03187207 0.024% AM | PF-03187207 0.040% AM | PF-03187207 0.040% PM | Latanoprost 0.005% AM | Latanoprost 0.005% PM
Number analyzed (Participants) | 38 | 29 | 25 | 24 | 38
Participants | 1 | 1 | 3 | 0 | 2

ADVERSE EVENTS:
Time Frame: 28 days
Description: The safety population was utilized for adverse event summaries. The safety population included participants randomized with at least 1 dose of study medication; by treatment received even if randomized treatment assignment differed.
Arm/Group | PF-03187207 0.024% AM | PF-03187207 0.040% AM | PF-03187207 0.040% PM | Latanoprost 0.005% AM | Latanoprost 0.005% PM
Serious Adverse Events (participants affected / at risk) | 0/43 | 0/32 | 0/28 | 0/28 | 0/45
Other Adverse Events (participants affected / at risk) | 6/43 | 11/32 | 9/28 | 7/28 | 6/45
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PF-03187207 0.024% AM (N=43) | PF-03187207 0.040% AM (N=32) | PF-03187207 0.040% PM (N=28) | Latanoprost 0.005% AM (N=28) | Latanoprost 0.005% PM (N=45)
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 2 | 0 | 0
Conjunctival hyperaemia (Eye disorders) | 5 | 2 | 1 | 1 | 4
Eye irritation (Eye disorders) | 0 | 2 | 3 | 2 | 1
Eye pain (Eye disorders) | 0 | 3 | 1 | 1 | 0
Ocular hyperaemia (Eye disorders) | 1 | 1 | 2 | 0 | 1
Photophobia (Eye disorders) | 0 | 2 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 1 | 0 | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Contact sponsor directly for details.